CLINICAL TRIAL: NCT05766176
Title: Study of the Effectiveness of The COVID-19 Vaccine
Status: Completed | Type: Observational
Sponsor: Universitas Sebelas Maret (Other)
Responsible Party: Principal Investigator, Nurhasan Agung Prabowo, Head of Hospital Research Unit, Universitas Sebelas Maret
Other Study IDs: NAP04
Record Dates: First submitted 2023-03-09; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
Keywords: COVID-19 Vaccine, Health Worker
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Serological Testing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health worker: A health worker who received a second dose of booster COVID19 vaccine
  Interventions: Diagnostic Test: COVID-19 Antibody

INTERVENTIONS:
Diagnostic Test: COVID-19 Antibody — This descriptive study examines the levels of neutralizing antibodies against COVID-19 in health workers before and after the Quantitative Anti-SARS-CoV-2 Test is an examination to measure in vitro quantitative antibodies (including IgG) against the receptor binding domain (RBD) of the SARS-CoV Spike (S) protein. -2, which aims to assess the adaptive humoral immune response to the SARS-CoV-2 Spike protein. Measurement with the ECLIA method. Ratio Scale after the 2nd booster COVID-19 vaccine in Surakarta, Indonesia.
  Other Names: COVID-19 Immunoglobulin

SUMMARY:
This descriptive study examines neutralizing antibody levels against COVID-19 in health workers before and after the 2nd booster of the COVID-19 vaccine in Surakarta, Indonesia.

DETAILED DESCRIPTION:
This research is a cross-sectional study with a descriptive-analytic design, community-based, of adults who live in Surakarta (age 18 years and over) using the Google form. The inclusion criteria were health workers receiving the third or second dose of the COVID-19 vaccine. Quantitative antibody titers are checked at Prodia's laboratory. Other variables examined were the number and date of vaccination, age, sex, comorbid diseases, body mass index, AEFI symptoms after the vaccine, and history of being infected with COVID-19. In the statistical analysis using the different and regression correlation tests, the significance level of P is less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Health workers who receive the second booster of COVID-19 vaccination

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Health worker in Universitas Sebelas Maret Hospital, Surakarta, Indonesia
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
quantitative anti-sars-cov-2 titers | Change of quantitative anti-sars-cov-2 titers before the second booster of vaccination COVID-19 and one month after
  The quantitative Anti-SARS-CoV-2 test is an examination to measure in vitro quantitative antibodies (including IgG) against the receptor binding domain (RBD) of the SARS-CoV-2 Spike protein (S) which aims to assess the adaptive humoral immune response to the SARS-CoV-2 Spike protein. Measurement with the ECLIA method. Ratio Scale

CONTACTS AND LOCATIONS:
Overall Officials: Nurhasan Agung Prabowo, MD, Principal Investigator — Universitas Sebelas Maret
Locations (1):
- Universitas Sebelas Maret Hospital, Sukoharjo, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pratama YS, Pradiptakirana R, Rachmah A, Prabowo NA. Autoimmune Thrombocytopenia in SLE and COVID-19. Eur J Case Rep Intern Med. 2021 Nov 3;8(11):002863. doi: 10.12890/2021_002863. eCollection 2021. PMID 34912736
- [Result] Sholihah MM, Kusuma TRH, Hanif MI, Prabowo NA. Letter to the Editor on Type 1 diabetes onset triggered by COVID-19. Acta Diabetol. 2021 Sep;58(9):1283-1284. doi: 10.1007/s00592-021-01761-3. Epub 2021 Jun 28. No abstract available. PMID 34181079